CLINICAL TRIAL: NCT05116748
Title: Safety and Immunogenicity of the SARS-CoV2 Vaccine in Solid Organ Transplantation (Lung and / or Liver) Adult Recipients
Brief Title: COVID19 Vaccine in SOT Adult Recipients
Acronym: COVID19_VaxSOT
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Letizia Morlacchi, Principal Investigator; Respiratory Consultant, attending Lung Transplant clinic, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: COVID19_VaxSOT
Record Dates: First submitted 2021-09-28; First posted 2021-11-11 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Vaccine Adverse Reaction; Vaccine Response Impaired; Vaccine Reaction; Lung Transplant; Complications; Liver Transplant; Complications; Vaccination
Keywords: COVID19; Vaccination; Vaccine; Transplant; Solid organ transplant; Lung transplant; Liver transplant
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LuTx recipients: Lung Transplant recipients
  Interventions: Biological: COVID19 mRNA vaccine
- OLT recipients: Orthotopic Liver Transplant recipients
  Interventions: Biological: COVID19 mRNA vaccine

INTERVENTIONS:
Biological: COVID19 mRNA vaccine — Administration of COVID19 mRNA vaccine

SUMMARY:
Background: ISHLT and AASLD guidelines recommend SARS-CoV2 vaccination in all individuals undergoing lung and liver transplantation, but there are currently scarce data on the safety and efficacy of these vaccines in this population. In Italy, immunocompromised patients have received the indication to be administered mRNA vaccines only.

Primary outcome: safety and reactogenicity Secondary outcomes: immunogenicity and prevention of COVID19

Visits and timepoints:

* T0: before first dose administration: visit and venous sampling to assess baseline COVID19 serum status
* Telephone calls to assess safety and reactogenicity 1 and 2 days after each dose of vaccination
* T21 or 28 (based on vaccine; mRNA BNT162b2 and mRNA-1273, respectively): visit, venous sampling to assess immunogenicity
* Follow up visits after 60, 120, 180 and 365 from T0: visit and venous sampling to assess immunogenicity

DETAILED DESCRIPTION:
Several studies indicate that solid organ transplant recipients are at increased risk of severe SARS-CoV2 disease (COVID19) and increased mortality from it (Pereira MR, AmJT 2020; Fernandez-Ruiz M, AmJT 2020; Kates OS, ClinInfectDis 2020).

Both ISHLT (International Society of Heart and Lung Transplantation) and AASLD (American Association for the Study of Liver Disease) guidelines recommend vaccination of all individuals undergoing lung and liver transplantation, starting from 3/6 months after transplantation.

In Italy, the Ministry of Health and the Italian Medicines Agency (AIFA) have established that immunosuppressed subjects following organ transplantation are worthy of vaccination with mRNA vaccines, since the latter are currently those with the greatest efficacy demonstrated among those approved in this country.

Within the Institution where this study will be conducted, patients undergoing lung and liver transplantation will be vaccinated, according to priority levels dictated by existing co-morbidities and by the time elapsed since transplantation, with the COMIRNATY mRNA vaccine (BNT162b2) administered according to the vaccination schedule of 2 doses at a distance of 21 days from each other or with the MODERNA vaccine (mRNA-1273) administered according to a vaccination schedule of 2 doses at a distance of 28 days from each other.

At present, no definitive data are available on the efficacy and the immunogenicity of anti-SARS-CoV-2 vaccines in solid organ transplant recipients, although the initial findings are reassuring. mRNA vaccines appear to be safe in the transplant population, and have not raised any concern at present about the possible onset of rejection or other serious adverse events in the first period after their administration (Boyarsky BJ, Transplantation 2021).

The primary objective of this study is to evaluate the safety and reactogenicity of antiSARS-CoV2 mRNA vaccines in SOT recipients.

Secondary outcomes include immunogenicity and efficacy (see Outcome paragraph for details).

Visits and timepoints:

* T0: before first dose administration: visit and venous sampling to assess baseline COVID19 serum status
* Telephone calls to assess safety and reactogenicity 1 and 2 days after each dose of vaccination
* T21 or 28 (based on vaccine; mRNA BNT162b2 and mRNA-1273, respectively): visit, venous sampling to assess immunogenicity
* Follow up visits after 60, 120, 180 and 365 from T0: visit and venous sampling to assess immunogenicity

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient's written informed consent

Exclusion Criteria:

* Lung transplant being performed in the previous 6 months
* Liver transplant being performed in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung and liver transplant recipients
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity | 365 days
  Primary endpoints:
  * Incidence of systemic and local adverse events (and their degree) in the subsequent 7 days after each vaccine administration in this population
  * Incidence of unusual adverse events (and their degree) in the subsequent 28 days after each vaccine administration in this population
  * Incidence of serious adverse events (SAEs) and sentinel events (NOCMCs, new onset chronic medical conditions, and MAAEs, medically-attended adverse events) over a 1-year follow-up period after administration of the first vaccine dose in this population

SECONDARY OUTCOMES:
Immunogenicity - antibody response, using ImmunoAssay in ECLIA for the quantitative detection of anti-protein S1 (spike) antibodies (including IgG) | 365 days
  * Geometric mean titer (GMT) of SARS-CoV2 anti-protein S1 total Ig (spike) antibody titers (GMT) at each timepoint
  * Percentage of individuals experiencing seroconversion at each timepoint
  * Increase of antibody titers (GMFR, geometric mean fold rise) from T0
Immunogenicity - Tcell response, using IGRA interferon-γ ELISpot, performed 60 days after the administration of the first vaccine dose | 60 days
  - Evaluation of the IFN-γ ELISpot-mediated T-cell response for different stimuli (peptides of proteins S1, S2, N, M, E and mix of structural proteins), measured with the following unit of measurement, i.e. IFN -γ spots / 250,000 PBMC (peripheral blood mononuclear cell) for each stimulus, 60 days after the first vaccine dose
Prevention of COVID19 | 365 days
  - Incidence of SARS-CoV2 infection, diagnosed with positivity of nasopharyngeal swab (SARS-CoV2 RNA search with RT-Real time PCR method)
Prevention of severe COVID19 | 365 days
  To evaluate the actual prevention of severe forms of SARS-CoV2 infection in this population
  - Incidence of severe forms of SARS-CoV2 infections, defined as requiring hospitalization of the patient and / or conditioning pneumonia / respiratory failure / sepsis / septic shock / ARDS
Immunogenicity and immunosuppression level | 365 days
  To compare the obtained (both antibody and T cell mediated) immunogenicity with the immunosuppression levels

CONTACTS AND LOCATIONS:
Overall Officials: Letizia Corinna Morlacchi, MD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Blumenthal KG, Robinson LB, Camargo CA Jr, Shenoy ES, Banerji A, Landman AB, Wickner P. Acute Allergic Reactions to mRNA COVID-19 Vaccines. JAMA. 2021 Apr 20;325(15):1562-1565. doi: 10.1001/jama.2021.3976. PMID 33683290
- [Background] Boyarsky BJ, Ou MT, Greenberg RS, Teles AT, Werbel WA, Avery RK, Massie AB, Segev DL, Garonzik-Wang JM. Safety of the First Dose of SARS-CoV-2 Vaccination in Solid Organ Transplant Recipients. Transplantation. 2021 May 1;105(5):e56-e57. doi: 10.1097/TP.0000000000003654. No abstract available. PMID 33560728
- [Background] Boyarsky BJ, Werbel WA, Avery RK, Tobian AAR, Massie AB, Segev DL, Garonzik-Wang JM. Immunogenicity of a Single Dose of SARS-CoV-2 Messenger RNA Vaccine in Solid Organ Transplant Recipients. JAMA. 2021 May 4;325(17):1784-1786. doi: 10.1001/jama.2021.4385. PMID 33720292
- [Background] Dagan N, Barda N, Kepten E, Miron O, Perchik S, Katz MA, Hernan MA, Lipsitch M, Reis B, Balicer RD. BNT162b2 mRNA Covid-19 Vaccine in a Nationwide Mass Vaccination Setting. N Engl J Med. 2021 Apr 15;384(15):1412-1423. doi: 10.1056/NEJMoa2101765. Epub 2021 Feb 24. PMID 33626250
- [Background] Fernandez-Ruiz M, Andres A, Loinaz C, Delgado JF, Lopez-Medrano F, San Juan R, Gonzalez E, Polanco N, Folgueira MD, Lalueza A, Lumbreras C, Aguado JM. COVID-19 in solid organ transplant recipients: A single-center case series from Spain. Am J Transplant. 2020 Jul;20(7):1849-1858. doi: 10.1111/ajt.15929. Epub 2020 May 10. PMID 32301155
- [Background] Fung M, Chiu CY, DeVoe C, Doernberg SB, Schwartz BS, Langelier C, Henrich TJ, Yokoe D, Davis J, Hays SR, Chandran S, Kukreja J, Ng D, Prostko J, Taylor R, Reyes K, Bainbridge E, Bond A, Chin-Hong P, Babik JM. Clinical outcomes and serologic response in solid organ transplant recipients with COVID-19: A case series from the United States. Am J Transplant. 2020 Nov;20(11):3225-3233. doi: 10.1111/ajt.16079. Epub 2020 Jul 17. PMID 32476258
- [Background] Grasselli G, Greco M, Zanella A, Albano G, Antonelli M, Bellani G, Bonanomi E, Cabrini L, Carlesso E, Castelli G, Cattaneo S, Cereda D, Colombo S, Coluccello A, Crescini G, Forastieri Molinari A, Foti G, Fumagalli R, Iotti GA, Langer T, Latronico N, Lorini FL, Mojoli F, Natalini G, Pessina CM, Ranieri VM, Rech R, Scudeller L, Rosano A, Storti E, Thompson BT, Tirani M, Villani PG, Pesenti A, Cecconi M; COVID-19 Lombardy ICU Network. Risk Factors Associated With Mortality Among Patients With COVID-19 in Intensive Care Units in Lombardy, Italy. JAMA Intern Med. 2020 Oct 1;180(10):1345-1355. doi: 10.1001/jamainternmed.2020.3539. PMID 32667669
- [Background] Kates OS, Haydel BM, Florman SS, Rana MM, Chaudhry ZS, Ramesh MS, Safa K, Kotton CN, Blumberg EA, Besharatian BD, Tanna SD, Ison MG, Malinis M, Azar MM, Rakita RM, Morilla JA, Majeed A, Sait AS, Spaggiari M, Hemmige V, Mehta SA, Neumann H, Badami A, Goldman JD, Lala A, Hemmersbach-Miller M, McCort ME, Bajrovic V, Ortiz-Bautista C, Friedman-Moraco R, Sehgal S, Lease ED, Fisher CE, Limaye AP; UW COVID-19 SOT Study Team. Coronavirus Disease 2019 in Solid Organ Transplant: A Multicenter Cohort Study. Clin Infect Dis. 2021 Dec 6;73(11):e4090-e4099. doi: 10.1093/cid/ciaa1097. PMID 32766815
- [Background] Long L, Zeng X, Zhang X, Xiao W, Guo E, Zhan W, Yang X, Li C, Wu C, Xu T, Zhan C, Chen Y, Jiang M, Zhong N, Lai K. Short-term outcomes of COVID-19 and risk factors for progression. Eur Respir J. 2020 May 27;55(5):2000990. doi: 10.1183/13993003.00990-2020. Print 2020 May. PMID 32312863
- [Background] Morlacchi LC, Rossetti V, Gigli L, Amati F, Rosso L, Aliberti S, Nosotti M, Blasi F. COVID-19 in lung transplant recipients: A case series from Milan, Italy. Transpl Infect Dis. 2020 Dec;22(6):e13356. doi: 10.1111/tid.13356. Epub 2020 Jun 26. PMID 32510771
- [Background] Pereira MR, Mohan S, Cohen DJ, Husain SA, Dube GK, Ratner LE, Arcasoy S, Aversa MM, Benvenuto LJ, Dadhania DM, Kapur S, Dove LM, Brown RS Jr, Rosenblatt RE, Samstein B, Uriel N, Farr MA, Satlin M, Small CB, Walsh TJ, Kodiyanplakkal RP, Miko BA, Aaron JG, Tsapepas DS, Emond JC, Verna EC. COVID-19 in solid organ transplant recipients: Initial report from the US epicenter. Am J Transplant. 2020 Jul;20(7):1800-1808. doi: 10.1111/ajt.15941. Epub 2020 May 10. PMID 32330343
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Sette A, Crotty S. Adaptive immunity to SARS-CoV-2 and COVID-19. Cell. 2021 Feb 18;184(4):861-880. doi: 10.1016/j.cell.2021.01.007. Epub 2021 Jan 12. PMID 33497610
- [Background] Shimabukuro TT, Cole M, Su JR. Reports of Anaphylaxis After Receipt of mRNA COVID-19 Vaccines in the US-December 14, 2020-January 18, 2021. JAMA. 2021 Mar 16;325(11):1101-1102. doi: 10.1001/jama.2021.1967. No abstract available. PMID 33576785
- [Background] Tschopp J, L'Huillier AG, Mombelli M, Mueller NJ, Khanna N, Garzoni C, Meloni D, Papadimitriou-Olivgeris M, Neofytos D, Hirsch HH, Schuurmans MM, Muller T, Berney T, Steiger J, Pascual M, Manuel O, van Delden C; Swiss Transplant Cohort Study (STCS). First experience of SARS-CoV-2 infections in solid organ transplant recipients in the Swiss Transplant Cohort Study. Am J Transplant. 2020 Oct;20(10):2876-2882. doi: 10.1111/ajt.16062. Epub 2020 Jun 9. PMID 32412159
- [Background] Xiang F, Wang X, He X, Peng Z, Yang B, Zhang J, Zhou Q, Ye H, Ma Y, Li H, Wei X, Cai P, Ma WL. Antibody Detection and Dynamic Characteristics in Patients With Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 5;71(8):1930-1934. doi: 10.1093/cid/ciaa461. PMID 32306047
- See also: Agenzia Italiana del Farmaco. — https://www.aifa.gov.it/vaccini-covid-19
- See also: Ministero della Salute del Governo Italiano — https://www.salute.gov.it/portale/home.html
- See also: Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/ctcae_v5_quick_reference_5x7.pdf
- See also: World Health Organization — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: NY Times vaccine tracker — https://www.nytimes.com/interactive/2020/science/coronavirus-vaccine-tracker.html